CLINICAL TRIAL: NCT02959177
Title: A Randomized, Double-Blind, Placebo-Controlled Study of LY2951742 (Galcanezumab) in Japanese Patients With Episodic Migraine
Brief Title: A Study of LY2951742 (Galcanezumab) in Japanese Participants With Episodic Migraine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15796; I5Q-JE-CGAN (Other: Eli Lilly and Company)
Record Dates: First submitted 2016-11-07; First posted 2016-11-08 (Estimated); Results first posted 2020-02-21 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2019-02

CONDITIONS: Migraine
Keywords: prevention; prophylaxis; headache
MeSH Terms: conditions — Migraine Disorders; Headache | interventions — galcanezumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 120 milligrams (mg) Galcanezumab (Experimental): 120 mg galcanezumab (LY2951742) administered subcutaneously (SC) once a month for 6 months.
  Interventions: Drug: Galcanezumab
- 240 mg Galcanezumab (Experimental): 120 mg galcanezumab (LY2951742) administered SC once a month for 6 months.
  Interventions: Drug: Galcanezumab
- Placebo (Placebo Comparator): Placebo administered SC once a month for 6 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Galcanezumab — Administered SC
  Other Names: LY2951742
  Arms: 120 milligrams (mg) Galcanezumab; 240 mg Galcanezumab
Drug: Placebo — Administered SC
  Arms: Placebo

SUMMARY:
The main purpose of this study is to determine the efficacy of the study drug Galcanezumab in Japanese participants with episodic migraine.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of migraine as defined by International Headache Society (IHS) International Classification of Headache Disorders (ICHD)-3 beta guidelines (1.1 or 1.2) (ICHD-3 2013), with a history of migraine headaches of at least 1 year prior to screening, and migraine onset prior to age 50.

Exclusion Criteria:

* Are currently enrolled in or have participated within the last 30 days or within 5 half-lives (whichever is longer) in a clinical trial involving an investigational product.
* Current use or prior exposure to Galcanezumab or other antibodies to CGRP or its receptor.
* Known hypersensitivity to multiple drugs, monoclonal antibodies or other therapeutic proteins, or to Galcanezumab and the excipients in the investigational product.
* History of persistent daily headache, cluster headache or migraine subtypes including hemiplegic (sporadic or familial) migraine, ophthalmoplegic migraine, and migraine with brainstem aura (basilar-type migraine) defined by IHS ICHD-3 beta.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 459 (Actual)
Dates: Start 2016-11-09 (Actual); Primary Completion 2019-01-18 (Actual); Study Completion 2019-01-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (41):
- Japan (41):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chiba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chofu-shi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fukui
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fukuoka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Higashioka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hiroshima
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Iruma-Gun
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kagoshima
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kasaoka-shi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kawasaki
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kobe
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Kobe
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kochi
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Kōchi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kyoto
  - "For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician.", Matsuyama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Matsuyama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Minatoku
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Minatoku
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Morioka
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Morioka
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Niigata
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nishinomiya
  - "For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician.", Nishinomiya
  - For additional information regarding investigative sites for this trial, contact 1-888-545-5972 Mon - Fri, 9 AM to 4 PM or 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time or speak with your personal physician., Nishinomiya
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Okayama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Osaka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ota-shi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ōita
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saijo-shi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saitama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sapporo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sendai
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shibuya-ku
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shinjuku-ku
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shizuoka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tachikawa-shi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tokyo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tōyama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Yamaguchi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Yamanashi

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
  .
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Takeshima T, Doi H, Ooba S, Tanji Y, Ozeki A, Komori M. Clinical Evaluation After Discontinuation of Galcanezumab in Japanese Patients with Episodic and Chronic Migraine: Analysis of a Randomized, Placebo-Controlled Trial and Open-label Extension Study. Neurol Ther. 2024 Jun;13(3):697-714. doi: 10.1007/s40120-024-00602-z. Epub 2024 Apr 6. PMID 38581615
- [Derived] Shibata M, Nihira A, Tanji Y, Ozeki A, Imagawa H, Komori M. Galcanezumab Efficacy Through the Dosing Interval in Japanese Patients with Episodic Migraine: Post Hoc Analysis of a Phase 2 Randomized Trial. Neurol Ther. 2023 Dec;12(6):2007-2019. doi: 10.1007/s40120-023-00534-0. Epub 2023 Sep 12. PMID 37698836
- [Derived] Igarashi H, Shibata M, Ozeki A, Matsumura T. Galcanezumab Effects on Migraine Severity and Symptoms in Japanese Patients with Episodic Migraine: Secondary Analysis of a Phase 2 Randomized Trial. Neurol Ther. 2023 Feb;12(1):73-87. doi: 10.1007/s40120-022-00410-3. Epub 2022 Oct 20. PMID 36266558
- [Derived] Igarashi H, Shibata M, Ozeki A, Day KA, Matsumura T. Early Onset and Maintenance Effect of Galcanezumab in Japanese Patients with Episodic Migraine. J Pain Res. 2021 Nov 16;14:3555-3564. doi: 10.2147/JPR.S326905. eCollection 2021. PMID 34815708
- [Derived] Tatsuoka Y, Takeshima T, Ozeki A, Matsumura T. Treatment Satisfaction of Galcanezumab in Japanese Patients with Episodic Migraine: A Phase 2 Randomized Controlled Study. Neurol Ther. 2021 Jun;10(1):265-278. doi: 10.1007/s40120-021-00236-5. Epub 2021 Apr 9. PMID 33835383
- [Derived] Shibata M, Nakamura T, Ozeki A, Ueda K, Nichols RM. Migraine-Specific Quality-of-Life Questionnaire (MSQ) Version 2.1 Score Improvement in Japanese Patients with Episodic Migraine by Galcanezumab Treatment: Japan Phase 2 Study. J Pain Res. 2020 Dec 31;13:3531-3538. doi: 10.2147/JPR.S287781. eCollection 2020. PMID 33408512

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were randomized to a Treatment Phase with double-blind treatment arms and then could enter a Follow-up Post Treatment Phase.
Groups:
- 120 mg Galcanezumab: Participants received loading dose of 240mg (2 injections of 120mg each) galcanezumab at first dosing visit followed by 120mg galcanezumab once a month for 5 months by subcutaneous (SC)injection.
- 240 mg Galcanezumab: Participants received 240 mg galcanezumab administered SC once a month for 6 months.
Period: Double-Blind Treatment Phase
Arm/Group | 120 mg Galcanezumab | 240 mg Galcanezumab | Placebo
Started | 115 | 114 | 230
Received at Least 1 Dose of Study Drug | 115 | 114 | 230
Completed | 104 | 111 | 225
Not Completed | 11 | 3 | 5
Not completed — Adverse Event | 5 | 2 | 0
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 0
Not completed — Withdrawal by Subject | 5 | 0 | 5
Period: Follow-up Post Treatment Phase
Arm/Group | 120 mg Galcanezumab | 240 mg Galcanezumab | Placebo
Started (Entered Post Treatment Phase) | 52 (Not all participants entered Post Treatment Follow-up Phase) | 52 (Not all participants entered Post Treatment Follow-up Phase) | 100 (Not all participants entered Post Treatment Follow-up Phase)
Completed | 51 | 51 | 98
Not Completed | 1 | 1 | 2
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least one dose of study drug.
Groups:
- 120 mg Galcanezumab: Participants received loading dose of 240mg (2 injections of 120mg each) galcanezumab at first dosing visit followed by 120mg galcanezumab once a month for 5 months by subcutaneous injection.
- Placebo: Participants were administered placebo SC once a month for 6 months..
- Total: Total of all reporting groups
Arm/Group | 120 mg Galcanezumab | 240 mg Galcanezumab | Placebo | Total
Number analyzed (Participants) | 115 | 114 | 230 | 459
Age, Customized [Count of Participants; unit: Participants]
  Less than 20 years old | 1 | 0 | 1 | 2
  Greater than 20 years old | 114 | 114 | 229 | 457
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 95 | 96 | 196 | 387
  Male | 20 | 18 | 34 | 72
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 115 | 114 | 230 | 459
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 115 | 114 | 230 | 459
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 115 | 114 | 230 | 459
Migraine Headache Days (MHD) per month [Mean (Standard Deviation); unit: days per month] — Migraine Headache Day (MHD): A calendar day on which a migraine headache or probable migraine headache occurred.
  days per month | 8.6 (2.8) | 9.0 (3.0) | 8.6 (3.0) | 8.8 (2.9)

OUTCOME MEASURES:

1. Primary Outcome: Overall Mean Change From Baseline in the Number of Monthly Migraine Headache Days (MHD)
Description: Migraine Headache Day (MHD):A calendar day on which a migraine headache or probable migraine headache occurred.
  Migraine Headache : A headache, with or without aura, of ≥30 minutes duration with both of the following required features (A and B):
  A) At least 2 of the following headache characteristics: Unilateral location; Pulsatile quality; Moderate or severe pain intensity; Aggravation by or causing avoidance of routine physical activity; AND B) During headache at least one of the following: Nausea and/or vomiting; Photophobia and phonophobia; The overall mean is derived from the average of months 1 to 6 from mixed model repeat measures (MMRM) model. Least Square Mean (LSMEAN) was calculated using MMRM models with fixed categorical effects of treatment, month, and treatment-by-month interaction, as well as the continuous, fixed covariates of baseline value and baseline-by-month interaction.
Time Frame: Baseline, Month 1 through Month 6
Population: All randomized participants who received at least one dose of study drug and had baseline and at least one post baseline value.
Measure: Least Squares Mean (95% Confidence Interval); unit: Days
Arm/Group | 120 mg Galcanezumab | 240 mg Galcanezumab | Placebo
Number analyzed (Participants) | 115 | 114 | 230
Days | -3.60 [-4.25 to -2.96] | -3.36 [-4.01 to -2.71] | -0.59 [-1.05 to -0.14]
Statistical Analysis 1: Comparison: 120 mg Galcanezumab vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean Difference = -3.01, 95% CI 2-sided [-3.80 to -2.22]
Statistical Analysis 2: Comparison: 240 mg Galcanezumab vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -2.7, 95% CI 2-sided [-3.53 to -1.94]

2. Secondary Outcome: Percentage of Participants With a 50% or Greater Reduction From Baseline in Monthly Migraine Headache Days
Description: Migraine Headache Day (MHD): A calendar day on which a migraine headache or probable migraine headache occurred. A 50% responder in a particular month is any participant who has a ≥50% reduction from baseline in the monthly number of migraine headache attacks in a 30-day interval. It is derived from the average of months 1 to 6 from generalized linear mixed model repeated measures. Mean percentages of participants were calculated with a generalized linear mixed model repeated measures method with treatment, month and treatment by month, and baseline MHD category as fixed factors.
Time Frame: Baseline, Month 1 through Month 6
Population: as for outcome 1
Measure: Mean (Standard Error); unit: percentage of participants
Arm/Group | 120 mg Galcanezumab | 240 mg Galcanezumab | Placebo
Number analyzed (Participants) | 115 | 114 | 230
percentage of participants | 49.8 (3.4) | 48.2 (3.5) | 20.3 (2.0)
Statistical Analysis 1: Comparison: 120 mg Galcanezumab vs Placebo; Test type: Superiority; Odds Ratio (OR) = 3.89, 95% CI 2-sided [2.71 to 5.57]
Statistical Analysis 2: Comparison: 240 mg Galcanezumab vs Placebo; Test type: Superiority; Odds Ratio (OR) = 3.664, 95% CI 2-sided [2.54 to 5.23]

3. Secondary Outcome: Percentage of Participants With a 75% or Greater Reduction From Baseline in Monthly Migraine Headache Days
Description: Migraine Headache Day (MHD): A calendar day on which a migraine headache or probable migraine headache occurred. A 75% responder in a particular month is any participant who has a ≥75% reduction from baseline in the monthly number of migraine headache attacks in a 30-day interval. It is derived from the average of months 1 to 6 from generalized linear mixed model repeated measures. Mean percentages of participants were calculated with a generalized linear mixed model repeated measures method with treatment, month and treatment by month, and baseline MHD category as fixed factors.
Time Frame: Baseline, Month 1 through Month 6
Population: as for outcome 1
Measure: Mean (Standard Error); unit: percentage of participants
Arm/Group | 120 mg Galcanezumab | 240 mg Galcanezumab | Placebo
Number analyzed (Participants) | 115 | 114 | 230
percentage of participants | 25.5 (2.8) | 25.0 (2.8) | 9.6 (1.3)
Statistical Analysis 1: Comparison: 120 mg Galcanezumab vs Placebo; Test type: Superiority; Odds Ratio (OR) = 3.24, 95% CI 2-sided [2.14 to 4.89]
Statistical Analysis 2: Comparison: 240 mg Galcanezumab vs Placebo; Test type: Superiority; Odds Ratio (OR) = 3.16, 95% CI 2-sided [2.08 to 4.80]

4. Secondary Outcome: Percentage of Participants With a 100% Reduction From Baseline in Monthly Migraine Headache Days
Description: Migraine Headache Day (MHD): A calendar day on which a migraine headache or probable migraine headache occurred. A 100% responder in a particular month is any participant who has a 100% reduction from baseline in the monthly number of migraine headache attacks in a 30-day interval. It is derived from the average of months 1 to 6 from generalized linear mixed model repeated measures. Mean percentages of participants were calculated with a generalized linear mixed model repeated measures method with treatment, month and treatment by month, and baseline MHD category as fixed factors.
Time Frame: Baseline, Month 1 through Month 6
Population: as for outcome 1
Measure: Mean (Standard Error); unit: percentage of participants
Arm/Group | 120 mg Galcanezumab | 240 mg Galcanezumab | Placebo
Number analyzed (Participants) | 115 | 114 | 230
percentage of participants | 9.0 (1.5) | 8.1 (1.5) | 2.8 (0.6)
Statistical Analysis 1: Comparison: 120 mg Galcanezumab vs Placebo; Test type: Superiority; Odds Ratio (OR) = 3.47, 95% CI 2-sided [2.03 to 5.93]
Statistical Analysis 2: Comparison: 240 mg Galcanezumab vs Placebo; Test type: Superiority; Odds Ratio (OR) = 3.13, 95% CI 2-sided [1.79 to 5.44]

5. Secondary Outcome: Overall Mean Change From Baseline on the Migraine-Specific Quality (MSQ) of Life Questionnaire
Description: MSQ version 2.1 is a health status instrument consists of 14 items addressing 3 domains:(1)Role Function-Restrictive (items 1-7);(2)Role Function- Preventive (items 8-11);&(3)Emotional Function (items 12-14).Response options range from "none of the time" (value 1) to "all of the time" (value 6), & are reverse-recoded (value 6 to 1) before the domain scores are calculated. Total raw scores for each domain is the sum of the final item value for all of the items in that domain. After total raw score is computed for each domain & total score, they are transformed to a 0-100 scale with higher scores indicating a better health status & a positive change in scores reflecting functional improvement. The overall mean is derived from the average of months 4 to 6 from MMRM model. LSMean was calculated using MMRM model with treatment, month, treatment by month, baseline by month and baseline MHD category as fixed factors.
Time Frame: Baseline, Month 4 through Month 6
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | 120 mg Galcanezumab | 240 mg Galcanezumab | Placebo
Number analyzed (Participants) | 112 | 112 | 228
units on a scale | 17.13 [15.10 to 19.15] | 15.91 [13.89 to 17.93] | 10.12 [8.70 to 11.55]
Statistical Analysis 1: Comparison: 120 mg Galcanezumab vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean difference = 7.00, 95% CI 2-sided [4.54 to 9.46]
Statistical Analysis 2: Comparison: 240 mg Galcanezumab vs Placebo; Test type: Superiority; p < 0.01, Mixed Models Analysis; Mean Difference (Final Values) = 5.79, 95% CI 2-sided [3.33 to 8.24]

6. Secondary Outcome: Overall Mean Change From Baseline in Number of Migraine Headache Days With Acute Medication Use
Description: Migraine Headache Day (MHD) with Acute Medication Use: Calendar days on which migraine or probable migraine occurs, requiring acute medication.
  The overall mean is derived from the average of months 1 to 6 from MMRM model. LSMean was calculated using MMRM model with treatment, month, treatment by month, baseline, baseline by month, and baseline MHD category as fixed effects.
Time Frame: Baseline, Month 1 through Month 6
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: MDHs with medication use
Arm/Group | 120 mg Galcanezumab | 240 mg Galcanezumab | Placebo
Number analyzed (Participants) | 115 | 114 | 230
MDHs with medication use | -3.02 [-3.60 to -2.43] | -2.81 [-3.40 to -2.23] | -0.12 [-0.53 to 0.30]
Statistical Analysis 1: Comparison: 120 mg Galcanezumab vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean difference = -2.90, 95% CI 2-sided [-3.61 to -2.19]
Statistical Analysis 2: Comparison: 240 mg Galcanezumab vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean difference = -2.70, 95% CI 2-sided [-3.41 to -1.99]

7. Secondary Outcome: Mean Change From Baseline in the Patient Global Impression of Severity (PGI-S) Score
Description: The PGI-S scale is a patient-rated instrument that measures patients own global impression of their illness severity. The patient was instructed as follows: "Considering migraine as a chronic condition, how would you rate your level of illness?" Response options were from 1 ("normal, not at all ill") to 7 ("extremely ill"). Mean is derived from the average of months 4 to 6 from MMRM model. Least square mean (LSM) was calculated using an MMRM model with treatment, month, treatment by month, baseline, baseline by month, and baseline MHD category as fixed effects.
Time Frame: Baseline, Month 4 through Month 6
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | 120 mg Galcanezumab | 240 mg Galcanezumab | Placebo
Number analyzed (Participants) | 112 | 112 | 228
units on a scale | -0.25 [-0.40 to -0.10] | -0.41 [-0.56 to -0.25] | -0.15 [-0.26 to -0.04]

8. Secondary Outcome: Overall Mean Change From Baseline in Headache Hours
Description: Headache Hours is calculated as the total number of headache hours on which a headache occurred. Overall mean is derived from the average of months 1 to 6 from MMRM model. LSMean was calculated using the MMRM model with treatment, month, treatment by month, baseline, baseline by month and baseline MHD category.
Time Frame: Baseline, Month 1 through Month 6
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: hours per month
Arm/Group | 120 mg Galcanezumab | 240 mg Galcanezumab | Placebo
Number analyzed (Participants) | 115 | 114 | 230
hours per month | -14.56 [-18.10 to -11.01] | -16.46 [-20.02 to -12.90] | -2.73 [-5.25 to -0.22]
Statistical Analysis 1: Comparison: 120 mg Galcanezumab vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean Difference = -11.82, 95% CI 2-sided [-16.14 to -7.51]
Statistical Analysis 2: Comparison: 240 mg Galcanezumab vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean difference = -13.73, 95% CI 2-sided [-18.05 to -9.40]

9. Secondary Outcome: Mean Change From Baseline on the Migraine Disability Assessment Test (MIDAS) Total Score
Description: The MIDAS is a participant-rated scale which was designed to quantify headache-related disability over a 3-month period. This instrument consists of five items that reflect the number of days reported as missing or with reduced productivity at work or home, and the number of days of missed social events. Each item has a numeric response range from 0 to 90 days, if days are missed from work or home they are not counted as days with reduced productivity at work or home. The numeric responses are summed to produce a total score ranging from 0 to 270, in which a higher value is indicative of more disability.
  LSMean was calculated using MMRM model with treatment, month, treatment by month, baseline, baseline by month, and baseline MHD category as fixed factors.
Time Frame: Baseline, Month 6
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | 120 mg Galcanezumab | 240 mg Galcanezumab | Placebo
Number analyzed (Participants) | 114 | 113 | 229
units on a scale | -7.06 [-9.67 to -4.44] | -5.13 [-7.69 to -2.58] | -2.16 [-3.96 to -0.36]
Statistical Analysis 1: Comparison: 120 mg Galcanezumab vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; LSMean Difference = -4.90, 95% CI 2-sided [-8.06 to -1.73]
Statistical Analysis 2: Comparison: 240 mg Galcanezumab vs Placebo; Test type: Superiority; p < .001, Mixed Models Analysis; LSMean Difference = -2.97, 95% CI 2-sided [-6.08 to 0.14]

10. Secondary Outcome: Percentage of Participants With Positive Responses on Patient Satisfaction With Medication Questionnaire-Modified (PSMQ-M)
Description: The PSMQ-M is a self-rated scale which measures participants level of satisfaction with study medication.The scale has been modified for use in this study, assessing 3 items related to the clinical trial treatment over the past 4 weeks: satisfaction, preference, and side effects. Satisfaction responses range from "very unsatisfied" to "very satisfied" with the current treatment. Preference compares the current study medication to previous medications, with responses from "much rather prefer my previous medication" to "much rather prefer the medication administered to me during the study"
Time Frame: Month 6
Population: All randomized participants who received at least one dose of study drug and had Month 6 PSMQ-M measurement.
Measure: Number; unit: percentage of participants
Arm/Group | 120 mg Galcanezumab | 240 mg Galcanezumab | Placebo
Number analyzed (Participants) | 104 | 111 | 225
percentage of participants
  Satisfaction: Very satisfied | 35.58 | 44.14 | 7.56
  Satisfaction: Somewhat satisfied | 26.92 | 23.42 | 27.11
  Side effects: Much less side effects | 35.58 | 28.83 | 24.89
  Side effects: Less side effects | 22.12 | 33.33 | 25.78
  Preference: Prefer study medication | 40.38 | 34.23 | 28.00
  Preference: Much Prefer study medication | 22.12 | 27.03 | 3.11

11. Secondary Outcome: Number of Participants With Suicidal Ideations Collected by Columbia - Suicide Severity Rating Scale (C-SSRS)
Description: C-SSRS captures the occurrence, severity, and frequency of suicide-related thoughts during the assessment period. The scale includes suggested questions to solicit the type of information needed to determine if a suicide-related thoughts occurred. Some questions are binary responses (yes/no) and some are on a scale of 1 (low severity) to 5 (high severity). Suicidal ideation (SI): a "yes" answer to any of 5 suicidal ideation questions: wish to be dead, non-specific active suicidal thoughts, active suicidal ideation with any methods without intent to act, active suicidal ideation with some intent to act without specific plan, active suicidal ideation with specific plan and intent
Time Frame: Month 1 through Month 6
Population: All randomized participants who received at least one dose of study drug and had at least one post baseline C-SSRS assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | 120 mg Galcanezumab | 240 mg Galcanezumab | Placebo
Number analyzed (Participants) | 115 | 114 | 230
Participants
  Wish to be dead | 1 | 0 | 0
  Non-specific active suicidal thoughts | 0 | 0 | 0
  Active SI with no intent | 0 | 0 | 0
  Active SI with some intent | 0 | 0 | 0
  Active SI with specific plan and intent | 0 | 0 | 0

12. Secondary Outcome: Number of Participants With Suicidal Behaviors Assessed by Columbia - Suicide Severity Rating Scale (C-SSRS)
Description: C -SSRS captures occurrence, severity, and frequency of suicide-related thoughts and behaviors. Suicidal behavior is defined as a "yes" answer to any of 5 suicidal behavior questions: preparatory acts or behavior, aborted attempt, interrupted attempt, actual attempt, and completed suicide. Suicidal ideation is defined as a "yes" answer to any one of 5 suicidal ideation questions: wish to be dead, and 4 different categories of active suicidal ideation.
Time Frame: Month 1 through Month 6
Population: All randomized participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | 120 mg Galcanezumab | 240 mg Galcanezumab | Placebo
Number analyzed (Participants) | 115 | 114 | 230
Participants
  Preparatory acts or behavior | 0 | 0 | 0
  Aborted attempt | 0 | 0 | 0
  Non-fatal suicide attempt | 0 | 0 | 0
  Completed suicide | 0 | 0 | 0

13. Secondary Outcome: Percentage of Participants Developing Anti-Drug Antibodies (ADA) to Galcanezumab
Description: Treatment emergent ADA will be defined as any of the following:
  * A negative baseline result and a positive post-baseline ADA result with a titer ≥20. This is also called treatment-induced ADA.
  * A positive baseline result and a positive post-baseline ADA result with a ≥4-fold increase in titers (for example, baseline titer of 10 increasing to ≥40 post-baseline). This is called treatment-boosted ADA.
Time Frame: Baseline through Month 6
Population: All randomized participants who received at least 1 dose of study drug and had evaluable immunogenicity data.
Measure: Number; unit: percentage of participants
Arm/Group | 120 mg Galcanezumab | 240 mg Galcanezumab | Placebo
Number analyzed (Participants) | 115 | 114 | 230
percentage of participants | 9.57 | 10.53 | 1.30

14. Secondary Outcome: Pharmacokinetics (PK): Serum Concentration of Galcanezumab
Description: Pharmacokinetics (PK): Serum Concentration of Galcanezumab
Time Frame: Month 6
Population: All randomized participants who received at least one dose of study drug and had measurable serum concentrations.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter
Arm/Group | 120 mg Galcanezumab | 240 mg Galcanezumab
Number analyzed (Participants) | 104 | 111
nanograms per milliliter | 20400 (7490) | 40600 (18400)

15. Secondary Outcome: Total Plasma Concentration of Calcitonin Gene-Related Peptide (CGRP)
Description: Total Plasma Concentration of Calcitonin Gene-Related Peptide (CGRP)
Time Frame: Month 6
Population: All randomized participants who received at least one dose of study drug and had measurable CGRP concentrations.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter
Arm/Group | 120 mg Galcanezumab | 240 mg Galcanezumab | Placebo
Number analyzed (Participants) | 104 | 110 | 25
nanograms per milliliter | 4.35 (1.25) | 5.40 (1.53) | 0.634 (1.36)

ADVERSE EVENTS:
Time Frame: 10 months
Description: All randomized participants who received at least 1 dose of study drug during treatment phase and remained in follow-up phase.
  Gender specific events only occurring in male or female participants have had the number of participants At Risk adjusted accordingly.
Groups:
- Treatment Phase Placebo: Participants were administered placebo SC once a month for 6 months.
- Treatment Phase 120 mg Galcanezumab: Participants received loading dose of 240mg (2 injections of 120mg each) galcanezumab at first doing visit followed by 120mg galcanezumab once a month for 5 months by subcutaneous injection.
- Treatment Phase 240 mg Galcanezumab: Participants received 240 mg galcanezumab administered SC once a month for 6 months.
- Follow-up Phase Placebo; Follow-up 120 mg Galcanezumab; Follow-up Phase 240 mg Galcanezumab: Participants did not receive study drug
Arm/Group | Treatment Phase Placebo | Treatment Phase 120 mg Galcanezumab | Treatment Phase 240 mg Galcanezumab | Follow-up Phase Placebo | Follow-up 120 mg Galcanezumab | Follow-up Phase 240 mg Galcanezumab
All-Cause Mortality (participants affected / at risk) | 0/230 | 0/115 | 0/114 | 0/100 | 0/52 | 0/52
Serious Adverse Events (participants affected / at risk) | 0/230 | 3/115 | 1/114 | 1/100 | 0/52 | 0/52
Other Adverse Events (participants affected / at risk) | 149/230 | 98/115 | 93/114 | 30/100 | 21/52 | 20/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Phase Placebo (N=230) | Treatment Phase 120 mg Galcanezumab (N=115) | Treatment Phase 240 mg Galcanezumab (N=114) | Follow-up Phase Placebo (N=100) | Follow-up 120 mg Galcanezumab (N=52) | Follow-up Phase 240 mg Galcanezumab (N=52)
Sudden hearing loss (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth impacted (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Treatment Phase Placebo (N=230) | Treatment Phase 120 mg Galcanezumab (N=115) | Treatment Phase 240 mg Galcanezumab (N=114) | Follow-up Phase Placebo (N=100) | Follow-up 120 mg Galcanezumab (N=52) | Follow-up Phase 240 mg Galcanezumab (N=52)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eustachian tube patulous (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eustachian tube stenosis (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meniere's disease (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Motion sickness (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sudden hearing loss (Ear and labyrinth disorders) | 0 (0) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Autoimmune thyroiditis (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Goitre (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenopia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chalazion (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctival hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Corneal disorder (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye pruritus (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Foreign body sensation in eyes (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glaucoma (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ocular hypertension (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 2 (3) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 8 (9) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
Abdominal wall haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Allergic stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Barrett's oesophagus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chapped lips (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cheilitis granulomatosa (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (3) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dental caries (Gastrointestinal disorders) | 5 (5) | 7 (8) | 5 (5) | 1 (1) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 7 (7) | 4 (6) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erosive duodenitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric polyps (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 4 (5) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis eosinophilic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingival swelling (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia oral (Gastrointestinal disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oroantral fistula (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periodontal disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tooth disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth impacted (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth loss (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 4 (5) | 5 (5) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hangover (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site bruising (General disorders) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site dermatitis (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Injection site discolouration (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site eczema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 5 (9) | 17 (46) | 31 (84) | 0 (0) | 0 (0) | 0 (0)
Injection site haemorrhage (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site induration (General disorders) | 1 (1) | 3 (5) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Injection site inflammation (General disorders) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site mass (General disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 3 (3) | 7 (9) | 8 (14) | 0 (0) | 0 (0) | 0 (0)
Injection site pruritus (General disorders) | 0 (0) | 10 (24) | 23 (59) | 0 (0) | 0 (0) | 0 (0)
Injection site rash (General disorders) | 2 (3) | 0 (0) | 3 (6) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site swelling (General disorders) | 3 (4) | 12 (22) | 12 (22) | 0 (0) | 0 (0) | 0 (0)
Injection site urticaria (General disorders) | 0 (0) | 1 (1) | 1 (4) | 0 (0) | 0 (0) | 0 (0)
Injection site warmth (General disorders) | 0 (0) | 2 (7) | 1 (4) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema (General disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Papillitis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Puncture site induration (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bacterial vulvovaginitis (Infections and infestations) | 0/196 (0) | 1/95 (1) | 0/96 (0) | 0/84 (0) | 0/43 (0) | 0/44 (0)
Bronchitis (Infections and infestations) | 1 (1) | 3 (3) | 1 (2) | 1 (1) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 2 (2) | 1 (1) | 3 (4) | 0 (0) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 5 (5) | 7 (7) | 3 (3) | 1 (1) | 3 (3) | 0 (0)
Gastroenteritis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Helicobacter infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hordeolum (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 3 (3) | 9 (10) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 76 (103) | 31 (43) | 28 (34) | 4 (5) | 4 (5) | 4 (5)
Oesophageal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 2 (3) | 2 (3) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Otitis externa (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pericoronitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periodontitis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 9 (9) | 4 (4) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulpitis dental (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 4 (5) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tinea pedis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urethritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvitis (Infections and infestations) | 0/196 (0) | 0/95 (0) | 1/96 (1) | 0/84 (0) | 0/43 (0) | 0/44 (0)
Vulvovaginal candidiasis (Infections and infestations) | 0/196 (0) | 0/95 (0) | 0/96 (0) | 0/84 (0) | 0/43 (0) | 1/44 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chillblains (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 4 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dental restoration failure (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Fractured coccyx (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fractured ischium (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Heat illness (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac function test abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Liver function test increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cells urine (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyslipidaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) | 6 (6) | 0 (0) | 1 (1) | 2 (2)
Fasciitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nodal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Kidney angiomyolipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cervical radiculopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Facial spasm (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intercostal neuralgia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Migraine with aura (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Migraine without aura (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 2 (2)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Occipital neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Poor quality sleep (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Radial nerve palsy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tension headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device failure (Product Issues) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neurosis (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast mass (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cervical dysplasia (Reproductive system and breast disorders) | 0/196 (0) | 0/95 (0) | 1/96 (1) | 0/84 (0) | 0/43 (0) | 0/44 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 1/196 (1) | 0/95 (0) | 1/96 (1) | 1/84 (2) | 0/43 (0) | 0/44 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0/196 (0) | 0/95 (0) | 0/96 (0) | 1/84 (1) | 0/43 (0) | 0/44 (0)
Premenstrual syndrome (Reproductive system and breast disorders) | 0/196 (0) | 0/95 (0) | 0/96 (0) | 1/84 (1) | 0/43 (0) | 0/44 (0)
Pruritus genital (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uterine polyp (Reproductive system and breast disorders) | 0/196 (0) | 1/95 (1) | 0/96 (0) | 0/84 (0) | 0/43 (0) | 0/44 (0)
Withdrawal bleed (Reproductive system and breast disorders) | 1/196 (1) | 0/95 (0) | 0/96 (0) | 0/84 (0) | 0/43 (0) | 0/44 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (4) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1) | 2 (5) | 0 (0) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alopecia areata (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asteatosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 2 (3) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hand dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rosacea (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin hypertrophy (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Solar dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3) | 7 (7) | 0 (0) | 0 (0) | 0 (0)
Xeroderma (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Menopause (Social circumstances) | 0 (0) | 0 (0) | 1 (1) | 0/84 (0) | 0/43 (0) | 0/44 (0)
Cyst removal (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Endodontic procedure (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Maxillary antrum operation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meniscus removal (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal septal operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin cyst excision (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tooth extraction (Surgical and medical procedures) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wisdom teeth removal (Surgical and medical procedures) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2016-08-30): https://cdn.clinicaltrials.gov/large-docs/77/NCT02959177/Prot_002.pdf
  • Statistical Analysis Plan (2018-11-15): https://cdn.clinicaltrials.gov/large-docs/77/NCT02959177/SAP_000.pdf